CLINICAL TRIAL: NCT02994641
Title: Critical Care Observation of Motor Activity (COMA) - A Practicable and Valid Predictor of Patients' Outcome in the Surgical Intensive Care Unit: A Observational Study at 2 Surgical Intensive Care Units at Massachusetts General Hospital
Brief Title: Critical Care Observation of Motor Activity (COMA) and SICU Outcomes
Acronym: COMA
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, Dr., Massachusetts General Hospital
Other Study IDs: 2015P002568
Record Dates: First submitted 2016-12-12; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Motor Activity; Muscle Strength; Muscle Weakness
Keywords: critical care; patient discharge; costs and cost analysis; length of stay; hospital mortality
MeSH Terms: conditions — Motor Activity; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adverse discharge disposition: Patients who were discharged to a skilled nursing facility or died in the hospital
  Interventions: Procedure: COMA Score Assessment
- No adverse discharge disposition: Patients who were not discharged to a skilled nursing facility or did not die in the hospital
  Interventions: Procedure: COMA Score Assessment

INTERVENTIONS:
Procedure: COMA Score Assessment

SUMMARY:
In the surgical intensive care unit (SICU), goals of critical care are often discussed in long-term ventilated patients around the time of extubation. Muscle weakness predicts extubation failure but formal muscle strength assessment by the Medical Research Council scale is time-consuming and not part of the daily clinical exam. In this observational study, we hypothesize that COMA measurement, routinely used by the SICU nurses, is a reliable and valid predictor for patients' SICU outcomes. This prospective observational study is carried out within a consecutively enrolled cohort of adult patients who are extubated in two SICUs at Massachusetts General Hospital, Boston.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated patients in 2 ICUs at Massachusetts General Hospital
* adult patients

Exclusion Criteria:

* Tracheostomy without extubation attempt
* Death without extubation attempt/terminal extubation

Ages: 18 Years to 112 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study cohort of adult patients who are extubated in two SICUs at Massachusetts General Hospital, Boston.
Sampling Method: Probability Sample
Enrollment: 761 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Adverse discharge disposition | Within one day after hospital discharge

SECONDARY OUTCOMES:
ICU length of stay | Time frame within 24 hours after ICU admission and within 24 hours after ICU discharge
Hospital length of stay | Time frame within 24 hours after hospital admission and within 24 hours after hospital discharge
30-day mortality | Within 30-days after extubation in the ICU or until the day of hospital discharge
Hospital costs | Between the day of hospital admission and the day of hospital discharge
30-day hospital readmission | Within 30 days after discharge from the index hospital stay

OTHER OUTCOMES:
Validation: Receiver operating curve (ROC) analysis - Acute Physiology and Chronic Health Evaluation II | At the day of admission to the ICU as well as within 72 hours after extubation
  ROC curve of COMA compared to ROC curve of Acute Physiology and Chronic Health Evaluation (APACHE) II
Validation: Receiver operating curve (ROC) analysis - Charlson Comorbidity Index | At the day of admission to the ICU as well as within 72 hours after extubation
  ROC curve of COMA compared to ROC curve of Charlson Comorbidity Index (CCI)
Validation: Receiver operating curve (ROC) analysis - Richmond Agitation and Sedation Score | Within 72 hours after extubation
  ROC curve of COMA compared to ROC curve of Richmond Agitation and Sedation Score (RASS)
Validation: Receiver operating curve (ROC) analysis - Confusion Assessment Method ICU score | Within 72 hours after extubation
  ROC curve of COMA compared to ROC curve of Confusion Assessment Method (CAM) ICU score
Validation: weighed kappa statistics | Within 72 hours after extubation
  Inter-rater agreement with COMA score between A.M. and P.M. shift nurse
Validation: correlation between COMA and actual skeletal muscle index assessed by computer tomography | Within 72 hours after extubation
  Skeletal muscle index is measured at the level of the 3rd lumbar vertebrae

CONTACTS AND LOCATIONS:
Locations (1):
- The Massachusetts General Hospital, Boston, Massachusetts, United States